CLINICAL TRIAL: NCT02999594
Title: Tramadol for Labor Analgesia in Low Risk Women: A Placebo Controlled Randomized Trial
Brief Title: Tramadol for Labor Analgesia: a Placebo Controlled Randomised Control Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Principal Investigator, dr aastha raheja, post graduate 1st year student obstetrics and gynecology department, Maulana Azad Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: mamc123
Record Dates: First submitted 2016-12-02; First posted 2016-12-21 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Tramadol for Labor Analgesia
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tramadol (Experimental): 50mg tramadol hydrochloride will be used intramuscularly as an experimental drug for evaluating its safety and efficacy as labor analgesic
  Interventions: Drug: Tramadol Hydrochloride
- distilled water (Placebo Comparator): 2ml distilled water intramuscularly will be used as a placebo.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Tramadol Hydrochloride — 50mg intramuscularly
  Arms: tramadol
Drug: Distilled Water — 2ml intramuscularly
  Arms: distilled water

SUMMARY:
Tramadol for labor analgesia: a low risk placebo controlled randomised control trial

DETAILED DESCRIPTION:
Investigators will administer 100mg tramadol or 2ml distilled water through intramuscular route in a blinded manner. Visual analogue score will be assessed in the beginning and every hour till four hours. patient satisfaction, safety outcomes, duration of 1st and 2nd stage of labor, proportion of women experiencing nausea, vomiting and increased sleepiness, postpartum haemorrhage,apgar score at 5 minute, need for nicu admission wiil be assessed at the end

ELIGIBILITY:
Inclusion Criteria:

* delivering for first time(nulliparous)
* well established labor ( 3 or more contractions in a span of ten minutes
* cervical dilation of 4 cm or more
* >= 80% effacement of cervix

Exclusion Criteria:

* any medical disorder- diabetes,hypertension
* obstetric high risk factors

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | at 2nd hour of administration
  visual analogue scale i.e scaling of severity of pain from 1 being mildest and 10 being most severe will be assessed at 2nd hour of administration

SECONDARY OUTCOMES:
patient satisfaction | at the end of labor( within 12 hours)
  scale of 1-5 including highly satisfied, moderately satisfied ,it is ok ,not satisfied ,highly unsatisfied
fetal distress | during labor
  fetal tachycardia (heart rate more than 160) or fetal bradycardia (heart rate less than 100)
duration of 1st and 2nd stage of labor | 1st and 2nd stage
women with side effects like postpartum haemorrhage, nausea, vomiting and increased sleepiness | till the end of labor
  increased risk of postpartum haemorrhage, nausea , vomiting and sleepiness may be associated with use of tramadol
neonatal safety in terms of apgar score and nicu admission | apgar score at 0 and 5 min
need for caesarean section or instrumental delivery | during labor
  emergency caesarean section or need for forceps or vacuum application

CONTACTS AND LOCATIONS:
Overall Officials: dr aastha raheja, Principal Investigator — Maulana Azad Medical College